CLINICAL TRIAL: NCT05300295
Title: Evaluation of a Mentorship Program for Individuals With Autism Spectrum Disorder (ASD)
Brief Title: Mentorship Program for Individuals With Autism Spectrum Disorder (ASD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00003954
Record Dates: First submitted 2022-02-24; First posted 2022-03-29 (Actual); Results first posted 2022-10-21 (Actual); Last update posted 2022-10-21 (Actual); Status verified 2022-10

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism; Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mentoring Program (Experimental): The Autism Mentorship Program is a psychosocial intervention that pairs adults and adolescents with autism spectrum disorder (ASD) in one-to-one mentoring relationships. AMP involves weekly meetings in an afterschool setting and targets the socio-emotional health and social connectedness of adolescents and adults with ASD.
  Interventions: Behavioral: Mentoring Program

INTERVENTIONS:
Behavioral: Mentoring Program — The Autism Mentorship Program is a psychosocial intervention that pairs adults and adolescents with autism spectrum disorder (ASD) in one-to-one mentoring relationships. AMP involves weekly meetings in an afterschool setting and targets the socio-emotional health and social connectedness of adolescents and adults with ASD.
  Other Names: Autism Mentorship Program

SUMMARY:
The purpose of this pilot project is to evaluate the feasibility of a mentorship program for adolescents with autism spectrum disorder (ASD). Data will be collected from adolescents with ASD and their parents/guardians. Study findings will be used to inform further development of the mentoring program for individuals with ASD.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of autism spectrum disorder (ASD)
* Age 14-18
* Participants in the mentoring program.
* Participants must have fluent language and will speak and understand English.
* Participants must be able to commit to providing evaluation data.

Exclusion Criteria:

* Have an intellectual disability (IQ under 70)

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lindsey Weiler, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mentoring Program
Started | 13
Completed | 13
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Mentoring Program: Mentoring Program: UMN staff will engage participants, parents, and program staff in pre-, mid-, and post-program interviews, focus groups, and surveys. Furthermore, UMN staff will have access to program applications completed by participants and will receive weekly information from program staff regarding attendance and participant ratings of the weekly meetings
Arm/Group | Mentoring Program
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 13
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 6
  More than one race | 1
  Unknown or Not Reported | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Sessions Attended
Description: Median count of completed session visits
Time Frame: within 30 days of the intervention end, up to 10 months
Measure: Median (Standard Deviation); unit: sessions
Arm/Group | Mentoring Program
Number analyzed (Participants) | 13
sessions | 13 (2.58)

2. Primary Outcome: Participant Program Satisfaction Scores
Description: Average program satisfaction score; range = 1-5; higher scores are better
Time Frame: within 30 days of the intervention end, up to 10 months
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Mentoring Program
Number analyzed (Participants) | 9
scores on a scale | 3.56 (1.13)

3. Primary Outcome: Mentoring Relationship Quality
Description: Average quality of the mentoring relationship score; range = 1-5; higher scores are better
Time Frame: within 30 days of the intervention end, up to 10 months
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Mentoring Program
Number analyzed (Participants) | 9
scores on a scale | 4.12 (0.52)

4. Primary Outcome: Child Behavior Checklist Scores (Internalizing Subscale)
Description: Parent-completed assessment of child's internalizing behavior; T scores for the internalizing subscale range 0-100 with higher scores being worse
Time Frame: at pre-intervention (within 30 days of intervention start) and post-intervention (within 30 days of intervention end), up to 10 months
Population: Some participants did not complete this post-intervention assessment.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Mentoring Program
Number analyzed (Participants) | 13
T-score
  Pre-intervention | 60.92 (9.58)
  Post-intervention: number analyzed (Participants) | 10
  Post-intervention | 63.1 (7.91)

5. Primary Outcome: Child Behavior Checklist Scores (Externalizing Subscale)
Description: Parent-completed assessment of child's externalizing behavior; T scores for the externalizing subscale range 0-100 with higher scores being worse
Time Frame: as for outcome 4
Population: Some participants did not complete this post-intervention assessment.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Mentoring Program
Number analyzed (Participants) | 13
T-score
  Pre-intervention | 51.85 (9.15)
  Post-intervention: number analyzed (Participants) | 10
  Post-intervention | 55.3 (6.77)

6. Primary Outcome: Youth Self-Report Scores (Internalizing Subscale)
Description: Youth self-reported assessment of internalizing behavior; T scores for the internalizing subscale range 0-100 with higher scores being worse
Time Frame: as for outcome 4
Population: Some participants did not complete this post-intervention assessment.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Mentoring Program
Number analyzed (Participants) | 13
T-score
  Pre-intervention | 56.31 (11.94)
  Post-intervention: number analyzed (Participants) | 9
  Post-intervention | 52.44 (11.81)

7. Primary Outcome: Youth Self-Report Scores (Externalizing Subscale)
Description: Youth self-reported assessment of externalizing behavior; T scores for the externalizing subscale range 0-100 with higher scores being worse
Time Frame: as for outcome 4
Population: Some participants did not complete this post-intervention assessment.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Mentoring Program
Number analyzed (Participants) | 13
T-score
  Pre-intervention | 49.54 (9.55)
  Post-intervention: number analyzed (Participants) | 9
  Post-intervention | 48.33 (8.17)

8. Primary Outcome: Social Skills Improvement System Scores (Social Competence Scale; Parent-report)
Description: Parent-completed assessment of child's social competence; Standard scores for the social competence subscale range 40-160 with lower scores being worse
Time Frame: as for outcome 4
Population: Some participants did not complete this post-intervention assessment.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Mentoring Program
Number analyzed (Participants) | 13
Score on a scale
  Pre-intervention | 83.62 (14.56)
  Post-intervention: number analyzed (Participants) | 10
  Post-intervention | 85.5 (8.32)

9. Primary Outcome: Social Skills Improvement System Scores (Problem Behavior Scale; Parent-report)
Description: Parent-completed assessment of child's problem behavior; Standard scores for the problem behavior subscale range 40-160 with higher scores being worse
Time Frame: as for outcome 4
Population: Some participants did not complete this post-intervention assessment.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Mentoring Program
Number analyzed (Participants) | 13
Score on a scale
  Pre-intervention | 113.23 (12.52)
  Post-intervention: number analyzed (Participants) | 10
  Post-intervention | 118.0 (11.15)

10. Primary Outcome: Social Skills Improvement System Scores (Social Competence Scale; Youth-report)
Description: Youth self-reported assessment of social competence; Standard scores for the social competence subscale range 40-160 with lower scores being worse
Time Frame: as for outcome 4
Population: Some participants did not complete this post-intervention assessment.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Mentoring Program
Number analyzed (Participants) | 13
Score on a scale
  Pre-intervention | 95.0 (20.1)
  Post-intervention: number analyzed (Participants) | 10
  Post-intervention | 102.11 (13.3)

11. Primary Outcome: Social Skills Improvement System Scores (Problem Behavior Scale; Youth-report)
Description: Youth self-reported assessment of problem behavior; Standard scores for the problem behavior subscale range 40-160 with higher scores being worse
Time Frame: as for outcome 4
Population: Some participants did not complete this post-intervention assessment.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Mentoring Program
Number analyzed (Participants) | 13
Score on a scale
  Pre-intervention | 97.92 (10.67)
  Post-intervention: number analyzed (Participants) | 9
  Post-intervention | 101.78 (14.62)

ADVERSE EVENTS:
Time Frame: Baseline to study completion, up to 17 months
Arm/Group | Mentoring Program
All-Cause Mortality (participants affected / at risk) | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-09-09): https://cdn.clinicaltrials.gov/large-docs/95/NCT05300295/Prot_SAP_000.pdf
  • Informed Consent Form (2019-01-07): https://cdn.clinicaltrials.gov/large-docs/95/NCT05300295/ICF_001.pdf